CLINICAL TRIAL: NCT01641978
Title: Study of Interobserver Correlation of Glasgow Coma Scale in Critical Neurological Patients
Brief Title: Study of Glasgow Coma Scale in Neurological Patients
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Susana Arias Rivera, Graduada en Enfermería, Hospital Universitario Getafe
Other Study IDs: GLASGOW GETAFE
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-06

CONDITIONS: Individuality

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients: neurological level in critical patients

SUMMARY:
The assessment of the level of consciousness in patients admitted to intensive care units (ICU) can be complicated because the variables that are evaluated can be interpreted in a different way by different observers.

The main objective is to determine interobserver agreement of the Glasgow Coma Scale (GCS) among ICU nurses and assess whether professional experience change the results. Secondary objective: to determine interobserver agreement in each of the three components (motor response, verbal and eye opening) of the GCS

DETAILED DESCRIPTION:
Prospective observational study conducted in a multi-unit 18 beds, neurological and / or neurosurgical patients are included. Variables: Demographic, reason for admission, overall and its components GCS. The neurological assessment was performed by a minimum of 3 nurses. One of them applied algorithm and evaluation technique and all agreed independently valued response to stimuli. Interobserver agreement measured by the intraclass correlation coefficient (ICC) with confidence interval (CI) of 95%. This study was approved by the Ethics Committee of Clinical Trials hospital.

ELIGIBILITY:
Inclusion Criteria:

* neurologic patients

Exclusion Criteria:

* pregnants, under-ages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: neurologic patients
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susana Arias, RN, Principal Investigator — Hospital Universitario de Getafe
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: neurological and neurosurgical patients
Groups:
- Neurologic Level: Neurologic patients
Period: Overall Study
Arm/Group | Neurologic Level
Started | 125
Completed | 125
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neurologic Level
Number analyzed (Participants) | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 67
  >=65 years | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 82
Region of Enrollment [Number; unit: participants]
  Spain | 125

OUTCOME MEASURES:

1. Primary Outcome: Interobserver Correlation
Description: interobserver agreement of the Glasgow Coma Scale (GCS) among ICU nurses measured by the intraclass correlation coefficient (ICC) with confidence interval (CI) 95%
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of correlation
Arm/Group | Neurologic Level
Number analyzed (Participants) | 125
percentage of correlation | 98.9 [98.5 to 99.2]

2. Secondary Outcome: Severity in Glasgow Coma Scale (GCS) by Groups.
Description: The Glasgow Coma Scale is divided into three components which are scored separately: ocular response (assessment 1-4 points), motor response (assessment 1-6 points) verbal response (evaluation of 1-5 points).
  Scores for each component are added together to get the total that will range between a minimum of 3 points (which corresponds to a patient who does not open his eyes and no motor response to stimulation or verbal response) and a maximum value of 15 points (corresponding to a patient with open eyes, obeying orders and maintaining a consistent language).
  It has been considered that the GCS score between 15 and 13 points corresponds to a slight alteration of consciousness, a score of 12-9 points with moderate impairment and 8 points or less with a serious deterioration in level of consciousness.
Time Frame: 1 year
Population: Neurological and/or neurosurgical patients in ICU
Measure: Number (95% Confidence Interval); unit: percentage of correlation
Groups:
- Severe: patients with GCS < 9 points
- Moderate: patients with GCS 9 - 12 points
- Slight: patients with GCS > 12 points
Arm/Group | Severe | Moderate | Slight
Number analyzed (Participants) | 53 | 39 | 33
percentage of correlation | 95.0 [91.9 to 96.1] | 60.3 [31.0 to 78.4] | 90.3 [81.8 to 95.2]

3. Secondary Outcome: Years of Professional Experience for Nurses in Critical Care
Description: Influence of professional experience in the evaluation of neurological patients
Time Frame: 1 year
Population: Nurses with a minimum experience of three years in intensive care
Measure: Median (Inter-Quartile Range); unit: years
Groups:
- Critical Care Time Experience: Influence of work experience in the evaluation of neurological patients
Arm/Group | Critical Care Time Experience
Number analyzed (Participants) | 6
years | 14 [3 to 17]

ADVERSE EVENTS:
Time Frame: six months
Arm/Group | Neurologic Level
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes